CLINICAL TRIAL: NCT06407128
Title: Valvular Microbiota and Valvulopathy
Acronym: MICROVALV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RC31/22/0108
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Valvulopathy
Keywords: Microbiota
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collection of biological samples (Experimental): The samples (1ml blood sample + approximately 90-100mg of valve tissue + saliva, periodontal and feces samples) will be collected at the time of T0 inclusion in the cardiovascular surgery department.
  Interventions: Biological: Collection of biological samples

INTERVENTIONS:
Biological: Collection of biological samples — Collection of biological samples (blood sample + valve tissue sample + saliva, periodontal and feces sample)

SUMMARY:
Few teams in the world can reliably analyze tissue microbiota. In this regard, the present group has unique expertise in the analysis of blood and tissue microbiota, the first to describe in 2011.

Having a blood biomarker of this valve microbiota could help guide the therapeutic strategy before and after the intervention. This study will be the first to test the hypothesis that the analysis of the blood microbiota makes it possible to detect the carriage of a tissue microbiota in patients undergoing aortic valve replacement (AVR) for degenerative aortic valve disease and should also lay the foundations for a prospective study. intended to evaluate the impact of the blood and valve microbiota on the post-operative prognosis of these patients and the complications at one year. This would be a first proof of concept of the role of the tissue microbiota in valvular degeneration linked to aging.

ELIGIBILITY:
Inclusion Criteria:

* Indication for surgical AVR:

  * Tight RA:

    * symptomatic (dyspnea, syncope/lipothymia, angina);
    * and/or echocardiographic criterion:
* valve surface < 1cm2 (and/or 0.6cm2/m2);
* average transvalvular gradient > 40mmHg;
* aortic jet velocity (Vmax) > 4.0m/s;

  * or low transvalvular gradient (mean gradient < 40mmHg) + left ventricular ejection fraction (LVEF) < 50% but contractile reserve;
  * and/or high calcium score on CT angiography;

    * Asymptomatic tight RA and:
  * LVEF < 50% without other cause;
  * and/or symptoms during exercise;
  * and/or low surgical risk + severity criteria: Vmax > 5.5m/s (or progression > 0.3m/s/year), NT-proBNP level > 3Xnormal, severe pulmonary arterial hypertension (pulmonary systolic pressure > 60mmHg);

    * Moderate AR + concomitant surgical indication for another heart disease;
    * Severe AI: regurgitant orifice > 30mm2, regurgitated volume > 60ml/beat,
  * symptomatic (dyspnea, syncope/lipothymia, angina);
  * and/or left ventricular dysfunction: LVEF < 50%, end-diastolic diameter > 70mm, end-systolic diameter > 50mm (or > 25mm/m2);
  * and/or concomitant surgical indication for another heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of blood and tissue microbiota | 12 months
  Detection of a blood microbiota in the pre-operative sample and a valve microbiota in the operating part.

CONTACTS AND LOCATIONS:
Overall Officials: Jean PORTERIE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No